CLINICAL TRIAL: NCT06732336
Title: HER2-PET Imaging Using 89Zr-trastuzumab in Low HER2-expressing (HER2-low) Breast Cancers
Brief Title: HER2-PET Imaging in HER2-low Breast Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-5574
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Metastatic
Keywords: HER2; HER2-low; PET; Breast cancer; 89Zr-trastuzumab
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 89Zr-trastuzumab PET imaging of HER2-low breast cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-trastuzumab PET/CT imaging of HER2-low patients (Experimental): Following their inform consent, HER2-low breast cancer patients will be invited to come to our research center twice. The first time patients will receive an intravenous dose of 10-50mg trastuzumab, followed by a 0.5 MBq/kg (max 60 MBq) dose of 89Zr-trastuzumab. Patients will come back for a second visit 3-6 days later to get their PET/CT imaging examination. Images will be evaluated by two PET-trained physicians, and analysed by an imaging scientist.
  Interventions: Diagnostic Test: 89Zr-trastuzumab

INTERVENTIONS:
Diagnostic Test: 89Zr-trastuzumab — Patients will receive an intravenous dose of 0.5 MBq/kg (max 60 MBq) of 89Zr-trastuzumab in order to perform a PET imaging session 3-6 days later.

SUMMARY:
A strategy to target the oncogenic receptor HER2 using a version of the anti-HER2 therapeutic antibody trastuzumab coupled to desferrioxamine (DFO) and radiolabeled with zirconium-89 ([89Zr]-DFO-trastuzumab) has been successfully evaluated in our group in preclinical settings. Clinical studies by other groups in recent years have shown the potential of targeting HER2+ lesions with [89Zr]-DFO-trastuzumab in patients with HER2+ cancers. We now want to establish the diagnostic potential of a protocol adding [89Zr]-DFO-trastuzumab PET imaging to FDG PET already used in the clinic for the detection of HER2-expressing cancers, including low expression levels considered until now as HER2-negative (HER2-low, IHC score 1+ and 2+ without FISH amplification of the HER2 locus). The HER2-low status has recently gained relevance thanks to large studies showing the efficacy of immunotherapy combined with drugs such as Enhertu (trastuzumab-deruxtecan), while trastuzumab alone was traditionally only effective for HER2+ cancers (IHC score 2+/FISH+, or 3+). In particular, we aim to develop a method to assess whole-body intertumoral heterogeneity in HER2 expression in order to detect cases with heterogeneous diseases and thus better stage patients and guide the optimal choice of personalized and targeted treatment to use. More specifically, the project aims to image with [89Zr]-DFO-trastuzumab PET patients with cancer, particularly breast cancer, but also esophageal, gastric, ovarian, endometrial and lung cancer, and whose primary tumor status is HER2-low.

DETAILED DESCRIPTION:
According to the Canadian Cancer Society, it is estimated that there were 28,600 new cases of breast cancer and 5,500 deaths due to the disease in Canada in 2022. Early stage, estrogen receptor-positive (ER+) tumor lesions are normally treated with resection, chemotherapy, and then hormone therapy and have the best prognosis for cure1. However, cases with metastases2, receptor-negative (ER-)3, and/or recurrence4 have a poor outcome and increased mortality. However, overexpression of the pro-oncogene Human Epithelial growth factor Receptor 2 (HER2), with or without ER expression, is linked to more aggressive cancers with poor prognoses5. Thus, ER and HER2 status are two of the most important prognostic factors for breast cancer and are routinely monitored on biopsy and tumor resection samples in pathology. HER2 status is also important to know in a range of cancers, including esophageal,6 gastric,7 ovarian,8 endometrial,9 and lung.10

However, it has been reported that in breast cancer patients with HER2 overexpression treated with a combination of chemotherapy and Herceptin (trastuzumab), a HER2-targeted antibody, the status of a potential recurrence will be HER2- in 43% of cases.11 A receptor status mismatch has been found between primary lesions and metastatic sites in 15% of patients for HER2 at initial workup.12-13 These data show that a substantial number of metastatic and/or recurrent breast cancers have heterogeneous disease, for which conventional primary and locoregional biopsy methods will fail to identify the optimal treatment plan and provide an accurate prognosis.

Although the feasibility of taking biopsies from suspected metastatic sites has been demonstrated to monitor the status of distal lesions14, it is difficult or impossible to take biopsy samples from all known and suspected sites for each patient, especially without knowing the precise metastatic status of each patient. This finding therefore highlights the need for a pan-body and non-invasive method of assessment and detection of HER2 for better cancer management and better use of targeted therapies.

Several medical imaging modalities allow the detection and monitoring of whole-body cancers. Among these, [18F]-fluorodeoxyglucose (FDG) positron emission tomography (PET) is routinely used for the initial assessment and staging16 as well as for monitoring of cancer treatment15, and this with high sensitivity and precision. On the other hand, FDG is not a tumor-specific tracer, and its uptake only reflects the relative avidity of a given tissue for glucose. Consequently, the physiological distribution and/or the presence of non-cancerous pathologies can reduce tumor contrast, even mask certain lesions, or lead to false positives17.

Trastuzumab and other antibodies targeting HER2 (Kadcyla, pertuzumab, etc.) are commonly used in the clinic and are very effective immunotherapies for the treatment of these very aggressive and previously very difficult to treat tumors. A few groups have already radiolabeled trastuzumab with zirconium-89 ([89Zr]-DFO-trastuzumab), and animal18 and human19 PET imaging studies have been successfully conducted. In 2016, the first data derived from PET imaging of human dosimetry and biodistribution of [89Zr]-DFO-trastuzumab were reported by an American group20,24. Recently, our research group has also succeeded in producing [89Zr]-DFO-trastuzumab with a better molar activity (~25 MBq/nmol) than that reported elsewhere so far21-22. A preclinical protocol of PET imaging with 4FMFES (an ER tracer) and [89Zr]-DFO-trastuzumab in succession on mice bearing ER+ and HER2+ tumors was developed, allowing the detection and identification with high contrast of lesions with different ER and HER2 status21-22. No side effects were detected during the preclinical procedures, indicating that the formulation is adequate. Building on these results and the expertise developed during these projects, we aim to transpose [89Zr]-DFO-trastuzumab PET imaging into the clinic during a phase II study on a cohort of patients with HER2-low cancer (IHC of HER 2 to 1+ or 2+ out of 3)25. More specifically, this imaging protocol aims to assess whole-body HER2 status26 and thus be able to detect cases with heterogeneous disease, in addition to standard locoregional biopsies. Thus, a clinical phase II focusing on the evaluation of a PET/CT protocol using [89Zr]-DFO-trastuzumab in succession to clinically prescribed FDG on patients will be conducted in order to produce the equivalent of a whole body biopsy of HER2 by imaging.

ELIGIBILITY:
Inclusion Criteria:

* HER2-low metastatic breast cancer;
* At least 18 years-old ;
* Able to stay in supine position for at least 30 minutes;
* Written inform consent.

Exclusion Criteria:

* Pregnancy or concomitant breast feeding;
* Hepatic disorders such as cirrhosis, hepatitis, or any other liver condition judged as significant by the treating physician and that could impair the biliary excretion of 89Zr-trastuzumab;
* Renal disorders considered significant by the treating physician and that could impair the normal elimination of 89Zr-trastuzumab;
* Known hypersensitivity or allergy to trastuzumab, desferrioxamine, or any constituents of 89Zr-trastuzumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate 89Zr-trastuzumab PET imaging in a HER2-low breast cancer patient cohort | 18 months
  Patients (n=40) will be injected with a dose of 89Zr-trastuzumab, then imaged by PET/CT 3-6 days later. Images will be analysed, and each suspect foci will have a region-of-interest (ROI) drawn on it. 89Zr-trastuzumab uptake in suspected tumors will be measured as a standard uptake value (SUV). SUVs will be compared with the pathological status and grade from the primary tumor and/or distant biopsied lesions (when available).

CONTACTS AND LOCATIONS:
Overall Officials: Éric E Turcotte, MD, FRCPC, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No